CLINICAL TRIAL: NCT02860208
Title: Follow-Up After Surgical Treatment of Peri-implantitis
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: olivier2
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Peri-Implantitis
Keywords: Peri-Implantitis; Surgical therapy; Follow-up; Supportive peri-implant therapy
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 3 years follow-up: all patients who received surgical treatment for peri-implantitis during a Randomized and Controlled Trial registered in ClinicalTrials.gov NCT NCT01857804
  Interventions: Procedure: 3 years follow-up

INTERVENTIONS:
Procedure: 3 years follow-up — Examination 3 years after surgical treatment of peri-implantitis

SUMMARY:
The objective of this prospective clinical study was to evaluate the 3-year outcomes of anti-infective surgical treatment of peri-implantitis when a regular supportive peri-implant therapy (SPIT) programme was followed.

DETAILED DESCRIPTION:
The patients enrolled in this prospective study all received surgical treatment for peri-implantitis at one of 2 treatment centres (specialist periodontal practice, Molndal and Gothenburg, Public Dental Health Services, Region Vastra Gotaland, Sweden) and were enrolled between October 2010 and December 2013.). All were treated by experienced periodontists.

Details of the peri-implantitis treatment protocol have been described in a previous publication reporting on the 12-month clinical and radiographic treatment outcomes, registered at ClinicalTrials.gov (NCT01857804) and approved by the Regional Ethical Committee, Gothenburg, Sweden (Dnr. 654-10).

ELIGIBILITY:
Inclusion Criteria:

* all patients who received surgical treatment for peri-implantitis for 3 years ago

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all patients who received surgical treatment for peri-implantitis during the RCT registered in ClinicalTrials.gov NCT NCT01857804
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in treatment success at 3 years post-op | baseline (1 year post-op) and 3 years post-op
  treatment success is defined by pocket closure, no bleeding on probing, bone loss ≤0.5 mm between baseline and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tord Berglundh, Professor, Study Chair — Department of Periodontology, Institute of Odontology, The sahlgrenska academy, University of Gothenburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanz M, Chapple IL; Working Group 4 of the VIII European Workshop on Periodontology. Clinical research on peri-implant diseases: consensus report of Working Group 4. J Clin Periodontol. 2012 Feb;39 Suppl 12:202-6. doi: 10.1111/j.1600-051X.2011.01837.x. PMID 22533957
- [Background] Carcuac O, Derks J, Charalampakis G, Abrahamsson I, Wennstrom J, Berglundh T. Adjunctive Systemic and Local Antimicrobial Therapy in the Surgical Treatment of Peri-implantitis: A Randomized Controlled Clinical Trial. J Dent Res. 2016 Jan;95(1):50-7. doi: 10.1177/0022034515601961. Epub 2015 Aug 18. PMID 26285807
- [Background] Heitz-Mayfield LJA, Salvi GE, Mombelli A, Loup PJ, Heitz F, Kruger E, Lang NP. Supportive peri-implant therapy following anti-infective surgical peri-implantitis treatment: 5-year survival and success. Clin Oral Implants Res. 2018 Jan;29(1):1-6. doi: 10.1111/clr.12910. Epub 2016 Jun 23. PMID 27335316
- [Background] Serino G, Turri A. Outcome of surgical treatment of peri-implantitis: results from a 2-year prospective clinical study in humans. Clin Oral Implants Res. 2011 Nov;22(11):1214-20. doi: 10.1111/j.1600-0501.2010.02098.x. Epub 2011 Feb 11. PMID 21309860
- [Background] Serino G, Turri A, Lang NP. Maintenance therapy in patients following the surgical treatment of peri-implantitis: a 5-year follow-up study. Clin Oral Implants Res. 2015 Aug;26(8):950-956. doi: 10.1111/clr.12418. Epub 2014 May 26. PMID 24861154
- [Background] Mettraux GR, Sculean A, Burgin WB, Salvi GE. Two-year clinical outcomes following non-surgical mechanical therapy of peri-implantitis with adjunctive diode laser application. Clin Oral Implants Res. 2016 Jul;27(7):845-9. doi: 10.1111/clr.12689. Epub 2015 Sep 16. PMID 26374080